CLINICAL TRIAL: NCT00930722
Title: ASSET (Acupil® Non Interventional Study For Evaluation Of Safety Effectiveness And Tolerability)
Brief Title: A Non Interventional Study To Asses The Safety, Effectiveness And Tolerability Of Quinapril (Acupil®) In An Indian Population
Acronym: ASSET
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A9061066
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Results first posted 2011-05-04 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: Quinapril non-interventional/observational study safety
MeSH Terms: conditions — Hypertension | interventions — Quinapril

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- quinapril: quinapril
  Interventions: Drug: quinapril

INTERVENTIONS:
Drug: quinapril — per label as non interventional study
  Other Names: Acupil®

SUMMARY:
This is a prospective, non-interventional, non comparative drug study. The efficacy of Quinapril in Asian population has been evaluated, but specifically in Indian patients the data is sparse. Data in a real world setting in a large population of Indian patients would shed more light on the safety, tolerability and effectiveness of Quinapril in the Indian population.

ELIGIBILITY:
Inclusion Criteria:

* Patients already on therapy with Acupil® for a minimum period of 4 weeks, Evidence of a personally signed and dated informed consent document

Exclusion Criteria:

* Patients having a Week 0 visit blood pressure reading of more than 180/110 mm of Hg will not be eligible to participate in the study.
* Women of child bearing age, not willing to use contraceptives, will not be eligible for the study
* Women using oral contraceptives will also not be included in the study
* Patients who have received any drug other than Acupil® as the first prescribed antihypertensive would not be eligible for enrollment into the trial
* Patients having any complication at Week 0 visit which would require more thorough investigations or who required more than one anti-hypertensive drug at the time of initiation of their therapy will not be included in the study
* Patients having any contraindications as per the LPD of Acupil®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 400 patients will be included in this non-interventional study. Only hypertensive subjects, over the age of 18 years, and who have already been receiving Acupil® for a minimum duration of 4 weeks will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- India (13):
  - Pfizer Investigational Site, Patna, Bihar
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Ahmedabad, Maharashtra
  - Pfizer Investigational Site, Nagpur, Maharashtra
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Delhi, New Delhi
  - Pfizer Investigational Site, Jaipur, Rajasthan
  - Pfizer Investigational Site, Chennai, Tamil Nadu
  - Pfizer Investigational Site, Madurai, Tamil Nadu
  - Pfizer Investigational Site, Trichy, Tamil Nadu
  - Pfizer Investigational Site, Kanpur, Uttar Pradesh
  - Pfizer Investigational Site, Kolkata, West Bengal

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9061066&StudyName=A%20Non%20Interventional%20Study%20To%20Asses%20The%20Safety%2C%20Effectiveness%20And%20Tolerability%20Of%20Quinapril%20%28Acupil%AE%29%20In%20An%20Indian%20Population

RESULTS

PARTICIPANT FLOW:
Groups:
- Quinapril: Quinapril, starting at a dose of 10 milligram (mg) up to 80 mg once per day orally in accordance with the locally approved prescribing information, in participants who had already been receiving Quinapril for a minimum duration of 4 weeks.
Period: Overall Study
Arm/Group | Quinapril
Started | 329
Completed | 302
Not Completed | 27
Not completed — Lost to Follow-up | 16
Not completed — No longer willing to participate | 9
Not completed — Study terminated by sponsor | 2

BASELINE CHARACTERISTICS:
Arm/Group | Quinapril
Number analyzed (Participants) | 329
Age Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 145
  Male | 184

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Any untoward medical occurrence in a participant who received study drug was considered an AE, without regard to possibility of causal relationship. Treatment-emergent adverse events (TEAE): those which occurred or worsened after baseline. An AE resulting in any of the following outcomes, or deemed to be significant for any other reason, was considered to be a SAE: death; initial or prolonged inpatient hospitalization; a life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline to Week 52
Population: Full analysis set (FAS) included participants who received at least 1 dose of study medication including those who took it before enrollment.
Measure: Number; unit: Participants
Arm/Group | Quinapril
Number analyzed (Participants) | 329
Participants
  Adverse events | 1
  Serious adverse events | 0

2. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) at Week 12
Description: Value at week 12 minus value at baseline.
Time Frame: Baseline and Week 12
Population: FAS included all participants who received at least 1 dose of study medication including those who took it before enrollment. Missing values were imputed by last-observation-carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Quinapril
Number analyzed (Participants) | 329
Millimeters of mercury (mmHg)
  Baseline | 142.16 (12.93)
  Change at Week 12 | -9.40 (11.18)

3. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) at Week 12
Description: Value at week 12 minus value at baseline.
Time Frame: Baseline and Week 12
Population: FAS included all participants who received at least 1 dose of study medication including those who took it before enrollment. Missing values were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Quinapril
Number analyzed (Participants) | 329
mmHg
  Baseline | 86.31 (6.71)
  Change at Week 12 | -3.93 (6.29)

4. Secondary Outcome: Change From Baseline in SBP at Week 52
Description: Value at week 52 minus value at baseline.
Time Frame: Baseline and Week 52
Population: The "full analysis set - follow up" (FAS-FU) included the subset of participants who had at least 1 additional BP measurement. This analysis was not conducted because only 2 participants were eligible for inclusion in the FAS-FU.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Quinapril
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in DBP at Week 52
Description: Value at week 52 minus value at baseline.
Time Frame: Baseline and Week 52
Population: The FAS-FU included the subset of participants who had at least 1 additional BP measurement. This analysis was not conducted because only 2 participants were eligible for inclusion in the FAS-FU.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Quinapril
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Pre-treatment in SBP at Week 0
Description: Value at Week 0 minus value at pre-treatment. Pre-treatment BP was the last BP recorded before taking study medication from retrospective data. If no such value was available, the earliest retrospective BP value from medical records was considered.
Time Frame: Pre-treatment and Week 0
Population: FAS included all participants who received at least 1 dose of study medication including those who took it before enrolment. Missing values were imputed by LOCF.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Quinapril
Number analyzed (Participants) | 329
mmHg
  Pre-treatment | 154.06 (13.50)
  Change at Week 0 | -12.49 (11.69)

7. Secondary Outcome: Change From Pre-treatment in DBP at Week 0
Description: as for outcome 6
Time Frame: Pre-treatment and Week 0
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Quinapril
Number analyzed (Participants) | 329
mmHg
  Pre-treatment | 92.82 (7.91)
  Change at Week 0 | -6.74 (8.20)

8. Secondary Outcome: Number of Participants Achieving BP Goal at Week 12
Description: The status of achieving a participant's goal BP at Week 12 was yes (at goal) or no (not at goal). The BP goal also depended on the participant's status of "Diabetes Mellitus (DM) or renal disease". To be considered at goal, SBP/DBP must be less than 140/90 mmHg for participants without DM or renal disease and SBP/DBP must be less than 130/80 mmHg for participants with DM or renal disease.
Time Frame: Week 12
Population: FAS included all participants who received at least 1 dose of study medication including those who took it before enrolment. Subgroup analysis was performed for each subgroup of participants in the FAS defined by DM or renal disease status. Missing values were imputed by LOCF.
Measure: Number; unit: Participants
Arm/Group | Quinapril
Number analyzed (Participants) | 329
Participants | 78

9. Secondary Outcome: Number of Participants With Achievement of BP Goal at Week 52
Description: The status of achieving a participant's goal BP at week 52 was yes (at goal) or no (not at goal). The BP goal also depended on the participant's status of "DM or renal disease". To be considered at goal, SBP/DBP must be less than 140/90 mmHg for participants without DM or renal disease and SBP/DBP must be less than 130/80 mmHg for participants with DM or renal disease.
Time Frame: Week 52
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Quinapril
Number analyzed (Participants) | 0

10. Secondary Outcome: Duration of Monotherapy With Quinapril
Description: Time in weeks to the first "taking additional antihypertensive medication" since Quinapril therapy began.
Time Frame: Baseline up to week 52 or early termination
Population: FAS included all participants who received at least 1 dose of study medication including those who took it before enrollment. Missing values were not imputed. Due to limited number of participants available, the analysis could not be performed.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Quinapril
Number analyzed (Participants) | 0

11. Secondary Outcome: Mean Daily Dose of Study Medication
Description: The mean daily dose of the study medication was calculated by dividing the total dose (sum of the daily doses) in the study by the treatment duration.
Time Frame: Baseline up to week 52 or early termination
Population: FAS included all participants who received at least 1 dose of study medication including those who took it before enrollment. Missing values were not imputed.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Quinapril
Number analyzed (Participants) | 329
mg | 11.28 (3.06)

12. Secondary Outcome: Number of Participants With Preference for add-on Anti-hypertensive Therapy
Description: The first add-on antihypertensive therapy for each participant was the first additional antihypertensive medication since initiation of Quinapril. If the participant did not require any such add-on medication, the first add-on antihypertensive therapy was "None".
Time Frame: Baseline up to week 52 or early termination
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | Quinapril
Number analyzed (Participants) | 329
Participants
  None | 321
  Metoprolol | 1
  Metoprolol Succinate | 1

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Quinapril
Serious Adverse Events (participants affected / at risk) | 0/329
Other Adverse Events (participants affected / at risk) | 1/329
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Quinapril (N=329)
Abdominal pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.